CLINICAL TRIAL: NCT04199286
Title: Assessment of Symmetrical and Asymmetrical Horizontal Strabismus Surgery: Efficacy and Lateral Incomitance
Brief Title: Bilateral and Unilateral Horizontal Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minia University Hospital
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymmetrical surgery (Active Comparator): This asymmetrical horizontal muscle surgery done as recess-resect in one eye or 3 muscle surgery
  Interventions: Procedure: symmetrical and asymmetrical horizontal strabismus surgery
- Symmetrical (Active Comparator): This symmetrical horizontal muscle surgery includes bilateral medial rectus recession in esotropia cases or bilateral lateral rectus recession in exotropia
  Interventions: Procedure: symmetrical and asymmetrical horizontal strabismus surgery

INTERVENTIONS:
Procedure: symmetrical and asymmetrical horizontal strabismus surgery — surgery was done on the medial rectus muscle on both eyes, lateral rectus muscle in both eyes or medial and lateral rectus muscle in one eye

SUMMARY:
This study was done in alternating strabismus patients to compare symmetrical muscle surgery and asymmetrical one as regard efficacy and lateral incomitance after surgery

ELIGIBILITY:
Inclusion Criteria:

* more than 3 years old.
* alternating esotropia or exotropia

Exclusion Criteria:

* unilateral strabismus
* paralytic or restrictive strabismus

Ages: 4 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-21 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
There was 95% success rate in asymmetrical group compared with 90% in symmetrical one | one and half year
  This result was measured by simultaneous prism cover test and expressed in prism diopter

CONTACTS AND LOCATIONS:
Overall Officials: Sahar TA Abdelaziz, MD, Principal Investigator — Assistant professor
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Minya, Minya Governorate
  - Mohamed F K Ibrahiem, Minya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ismail AA, Abdelkader MF, Mohamed AA, Abdelaziz ST. Evaluation of Efficacy and Lateral Gaze Incomitance in Symmetrical and Asymmetrical Surgery for Concomitant Esotropia and Exotropia. Clin Ophthalmol. 2021 Aug 26;15:3613-3621. doi: 10.2147/OPTH.S326659. eCollection 2021. PMID 34471346